CLINICAL TRIAL: NCT04689152
Title: A Multicenter, Randomized, Open-label Phase III Clinical Trial to Evaluate Efficacy and Safety of the Cellgram-LC in Patients With Alcoholic Liver Cirrhosis
Brief Title: Clinical Trial to Evaluate the Efficacy and Safety of Cellgram-LC Administration in Patients With Alcoholic Cirrhosis
Acronym: Cellgram-LC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Pharmicell Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PMC-P-07
Record Dates: First submitted 2020-12-21; First posted 2020-12-30 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Alcoholic Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis, Alcoholic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Best Supportive care
- Injection group: Cellgram-LC (Experimental): Within 1 month after extracting bone marrow, directly inject 7X10^7 autologous bone marrow-derived mesenchymal stem cells within liver through the hepatic artery.
  Interventions: Biological: Cellgram-LC

INTERVENTIONS:
Biological: Cellgram-LC — Patients will receive single injection of Cellgram-LC(mesenchymal stem cell) hepatic artery.
  Other Names: Autologous bone marrow-derived mesenchymal stem cell
  Arms: Injection group: Cellgram-LC

SUMMARY:
This phase III clinical trial is designed to evaluate the efficacy and safety of autologous Mesenchymal Stem Cells (MSC) injected hepatic artery.

DETAILED DESCRIPTION:
To evaluate the efficacy and efficacy for 60 months after a single dose of Cellgram-LC in patients with alcoholic liver cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

1. At the time of screening, 19 or 70 years
2. Patients diagnosed with alcoholic cirrhosis by combining alcohol history, imaging and pathological examination results, and clinical symptoms at screening, and belonging to Child-Pugh grade B or C (Child-Pugh score of 7 or more)
3. Those whose survival period is more than 1 year when judged by the tester
4. Those who can perform hepatic artery catheterization by inserting a catheter into the hepatic artery at the judgment of the examiner
5. In the case of women of childbearing potential, a person who was confirmed negative in the pregnancy test at screening and agreed to use contraception* by the method permitted for this clinical trial during the clinical trial
6. Those who can conduct clinical trials according to the clinical trial protocol
7. A person who has consented in writing to voluntarily participate in this clinical trial

Exclusion Criteria:

1. Those with a history of solid cancer including Hepatocellular Carcinoma (HCC) (within 5 years before screening), those who have been diagnosed with solid cancer and are currently undergoing chemotherapy or those whose hepatocellular carcinoma has been confirmed by screening tests
2. Patients who underwent portal systemic shunting in the jugular vein
3. Patients with alcohol consumption or hepatotoxic drugs within 6 months prior to screening
4. Persons taking high-dose steroids, immunosuppressants, or antimicrobials due to severe infections for at least 1 month of screening
5. Those who have major surgical operations, long-term biopsy, or significant trauma as judged by the investigator within 3 months before screening
6. Those whose history of gastrointestinal bleeding is confirmed within 10 days of screening
7. Those whose medical history or accompanying diseases following the screening time is confirmed

   * If you have not been diagnosed with a malignant blood disease (acute myelogenous leukemia, acute lymphocytic leukemia, non-Hodgkins lymphoma, Hodgkins lymphoma, multiple myelopathy)
   * Severe aplastic anemia
   * Liver transplant history
   * Liver diseases of other causes besides alcoholic cirrhosis: hepatitis B and C, autoimmune liver disease (primary cholangitis, primary sclerosing cholangitis and autoimmune hepatitis, etc.), weak liver toxicity, non-alcoholic fatty liver disease , NAFLD), Wilson's disease, iron excess, alpha-1-antitrypsin deficiency, etc.)
   * Extrahepatic biliary stenosis
   * Active portal vein or hepatic vein thrombosis
   * Heart failure or respiratory failure
   * Severe renal impairment (when the result of serum creatinine test exceeds 1.5 times the upper limit of normal)
   * Acute or chronic infection requiring systemic treatment
   * Severe coagulation disorder (if the tester judges it as a severe coagulation disorder or one of the following 1 to 3; 1. bleeding predisposition, 2. coagulation, 3. platelet≤50,000/mm3 and INR≥1.5)
8. serologic test result (HIV, HAV, HBV, HCV, Syphilis infection) positive factor
9. Patients unable to collect bone marrow due to bone marrow disease
10. Those with a history of gentamicin hypersensitivity reaction
11. Pregnant or lactating women
12. Those with substance abuse experience within 1 year before screening
13. Those who participated in other clinical trials within one month before screening and administered (or applied) clinical trial drugs (or medical devices)
14. Those who previously participated in clinical trials related to cell therapy
15. Patients judged to be inappropriate to participate in this clinical trial due to complications, etc., when judged by the investigator before screening or registration

Ages: 20 Years to 71 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-03-02 (Actual); Primary Completion 2027-08-02 (Estimated); Study Completion 2028-01-02 (Estimated)

PRIMARY OUTCOMES:
Transplant free survival (TFS) | For 3 years
  Transplant free survival (TFS), the median survival time and 95% confidence interval for each group were presented using the Kaplan-Meier method, and the difference in the survival distribution between the two groups was used as a Cox proportional hazards model corrected for stratification Black.

SECONDARY OUTCOMES:
Survival rate | month 24 and 36
  For the survival rate, the survival rate and 95% confidence interval at each time point are presented using the Kaplan-Meier method, and the difference in survival rate between the two groups is tested using the Z statistic.
Change amount of Child-Pugh score | week -6 and 0
  In order to compare the difference between groups in the amount of change in each evaluation variable at the time of visit after cell administration/best supportive therapy compared to the baseline value, covariance analysis (ANCOVA) is performed by setting the baseline time point and stratification factor as a correction variable for each evaluation variable.
  CP score was calculated using five factors: hepatic encephalopathy, prothrombin time, bilirubin, serum albumin, and ascites, and the score range was 5-15 points.
  In the Child-Pugh grade, scores of the five factors are summed and evaluated as A if it is less than 7 points, B if it is 7-9, and C if it exceeds 9 points.
Change amount of MELD score | week -6 and 0
  In order to compare the difference between groups in the amount of change in each evaluation variable at the time of visit after cell administration/best supportive therapy compared to the baseline value, covariance analysis (ANCOVA) is performed by setting the baseline time point and stratification factor as a correction variable for each evaluation variable.
  The higher the score, the higher the mortality rate.
Change amount of Liver function test | month 0, 1, 3, 6, 9, 12, 18 and 24
  In order to compare the difference between groups in the amount of change in each evaluation variable at the time of visit after cell administration/best supportive therapy compared to the baseline value, covariance analysis (ANCOVA) is performed by setting the baseline time point and stratification factor as a correction variable for each evaluation variable.
Change amount of Fibrosis-4 | month 0, 6, 12, 18 and 24
  In order to compare the difference between groups in the amount of change in each evaluation variable at the time of visit after cell administration/best supportive therapy compared to the baseline value, covariance analysis (ANCOVA) is performed by setting the baseline time point and stratification factor as a correction variable for each evaluation variable.
Change amount of FibroScanⓇ | week -6 and 0
  In order to compare the difference between groups in the amount of change in each evaluation variable at the time of visit after cell administration/best supportive therapy compared to the baseline value, covariance analysis (ANCOVA) is performed by setting the baseline time point and stratification factor as a correction variable for each evaluation variable.
Change amount of EQ-5D | month -1, 6, 12, 18 and 24
  In order to compare the difference between groups in the amount of change in each evaluation variable at the time of visit after cell administration/best supportive therapy compared to the baseline value, covariance analysis (ANCOVA) is performed by setting the baseline time point and stratification factor as a correction variable for each evaluation variable.
  The higher the score, the higher the quality of life.
Change amount of EQ-VAS | month -1, 6, 12, 18 and 24
  In order to compare the difference between groups in the amount of change in each evaluation variable at the time of visit after cell administration/best supportive therapy compared to the baseline value, covariance analysis (ANCOVA) is performed by setting the baseline time point and stratification factor as a correction variable for each evaluation variable.
  The higher the score, the higher the quality of life.

OTHER OUTCOMES:
α-fetoprotein test | week -6, month 3, 6, 9, 12, 18, 24
  Two sample t-test or Wilcoxon rank-sum test is performed to test the difference between the two groups for the results of tumor marker test (AFP) at each time point.

CONTACTS AND LOCATIONS:
Overall Officials: Moonyoung Kim, Principal Investigator — Wonju Severance Christian Hospital
Locations (11):
- South Korea (11):
  - Soonchunhyang University Hospital, Bucheon-si
  - Soonchunhyang University Hospital, Cheonan
  - Gangwon National University Hospital, Chuncheon
  - Hallym Univ. Medical Center, Chuncheon
  - Gangneung Asan Hospital, Gangneung-si
  - Eunpyeong St. Mary's Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Soonchunhyang University Hospital, Seoul
  - Wonju Severance Christian Hospital, Wŏnju
  - Yongin Severance Hospital, Yŏngin